CLINICAL TRIAL: NCT05461222
Title: A Study of the Effectiveness of Fetal Endoscopic Tracheal Occlusion (FETO) in the Management of Severe Prenatally Diagnosed Congenital Diaphragmatic Hernia (CDH)
Brief Title: Fetal Endoscopic Tracheal Occlusion (FETO) for Severe Congenital Diaphragmatic Hernia
Acronym: FETO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yair Blumenfeld (Other)
Responsible Party: Sponsor-Investigator, Yair Blumenfeld, Associate Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 63230
Record Dates: First submitted 2022-07-13; First posted 2022-07-18 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Congenital Diaphragmatic Hernia
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Fetal Endoscopic Tracheal Occlusion (FETO) (Experimental): FETO is performed in-utero and the balloon is removed prior to delivery, and children will have follow-up visits until the age of 2
  Interventions: Device: Balt "Goldballoon"

INTERVENTIONS:
Device: Balt "Goldballoon" — Fetal endoscopic tracheal occlusion (FETO) is a procedure where a balloon is placed in the main airway or "windpipe" of the fetus, to help with the development of the lungs. This is performed using a fetoscope, a small camera that is inserted into the amniotic cavity and deploying the FETO Goldballoon into the fetal trachea.

SUMMARY:
The purpose of the study is to study the efficacy of fetal endoscopic tracheal occlusion (FETO) in cases of severe congenital diaphragmatic hernia (CDH). This study will also collect safety and effectiveness data for the off-label use of the FETO Goldballoon (the balloon that will be inserted into the fetal trachea), manufactured by Balt medical. The investigators hope to study the risks and benefits of FETO in cases of severe CDH in an advanced medical center such as Lucile Packard Children's Hospital (LPCH) Stanford with access to advanced maternal-fetal medicine, neonatal services, and neonatal ECMO, and pediatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Maternal Age: 18-50
* Singleton gestation
* Gestational age before 29 weeks 6 days
* Severe left or right-sided CDH: For severe left sided CDH observed-to-expected lung-to- head ratio (o/e LHR) less than 25% between 22 and 29 6/7 weeks' gestation, liver herniation, MRI lung volumes less than 30% expected based on gestational age nomograms. For severe right sided CDH o/e LHR less than 30 % between 22 and 29 6/7 weeks' gestation, liver herniation, MRI lung volumes less than 30% expected based on gestational age nomograms.
* Normal genetic karyotype or microarray testing by amniocentesis or chorionic villus sampling (CVS)
* Absence of associated fetal structural cardiac anomalies by a dedicated fetal echocardiogram
* Absence of other structural anomalies by ultrasound or MRI
* Appropriate multi-disciplinary counseling performed with maternal-fetal medicine, neonatology, pediatric surgery, genetics, pediatric otolaryngology (ENT).
* Must be willing to remain near LPCH Stanford (within 30 minutes from the hospital) for the duration of the balloon placement.
* No maternal and/or fetal contra-indications to fetal surgery such as a bleeding disorder, poorly controlled diabetes or hypertension, short cervix (measuring < 20mm), risk for preterm birth etc.
* Planned pregnancy surveillance at LPCH Stanford
* Planned delivery at LPCH Stanford
* Able to provide written consent
* Willingness to comply with all study procedures and availability (meets psychosocial criteria) for the duration of the study including having a support person

Exclusion Criteria:

* Contraindications to fetal surgery including poorly controlled hypertension, diabetes or other maternal medical condition including hematological disorder
* High risk for preterm labor and/or delivery based on either significant history of preterm birth, short cervix (measuring < 20mm), significant uterine anomaly or other risk factor, incompetent cervix (requiring cerclage)
* Non-isolated CDH - CDH with additional structural anomalies
* Significant maternal obesity defined as a body mass index (BMI) greater than 40. BMI is a calculation which includes a person's height and weight
* History of natural rubber latex allergy
* Uterine anomaly such as large or multiple fibroids or mullerian duct abnormality
* Participation in another intervention study that influences maternal and fetal morbidity and mortality.
* Bilateral CDH, left-sided CDH with O/E LHR >25%, or left-sided CDH with O/E LHR <25% but liver completely down in abdomen
* Right-sided CDH O/E LHR >30% or right-sided CDH with O/E LHR <30% with liver completely down in abdomen
* Significant placental abnormalities (abruption, chorioangioma, accreta) known at the time of enrollment and/or surgery
* Maternal-fetal Rhesus isoimmunization, Kell sensitization or neonatal alloimmune thrombocytopenia, affecting the current pregnancy.
* Maternal HIV, Hepatitis B with positive surface antigen, Hepatitis C with presence of virus in maternal blood due to risk of fetal transmission during the procedure
* No safe or feasible fetoscopic approach to balloon placement.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of neonates who survive until initial hospital discharge | Average approximately 6 months (up to 1 year)

SECONDARY OUTCOMES:
Number of neonates who survive until 28 days of life | 28 days
Number of children who survive until 6 months of age | 6 months
Number of children who survive until 1 year of age | 1 year
Number of children who survive until 2 years of age | 2 years
Number of children who receive extracorporeal membrane oxygenation (ECMO) | Average approximately 6 months (up to 1 year)

CONTACTS AND LOCATIONS:
Overall Officials: Yair Blumenfeld, MD, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No